CLINICAL TRIAL: NCT05189288
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-388 in Healthy Subjects
Brief Title: Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-388(2) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A99_03BE2122
Record Dates: First submitted 2022-01-02; First posted 2022-01-12 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-01

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference-Test (Experimental): D418 Tab. - CKD-388 Tab.
  Interventions: Drug: D418 Tab.; Drug: CKD-388 Tab.
- Test-Reference (Experimental): CKD-388 Tab. - D418 Tab.
  Interventions: Drug: D418 Tab.; Drug: CKD-388 Tab.

INTERVENTIONS:
Drug: D418 Tab. — 1T
  Other Names: Reference
Drug: CKD-388 Tab. — 1T
  Other Names: Test

SUMMARY:
This study is an open-label, randomized, single dose, crossover study to evaluate the pharmacokinetics, safety and tolerability of CKD-388 in healthy subjects

DETAILED DESCRIPTION:
To healthy 60 subjects, following treatments are administered dosing in each period and wash-out period is a minimum of 14 days.

Reference drug: D418 Tab. / Test drug: CKD-388 Tab. Pharmacokinetic blood samples are collected up to 72hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, aged ≥ 19 years old at the time of screening.
2. Weight ≥50kg (man) or 45kg (woman), with calculated body mass index (BMI) of 18 to 30 kg/m2 at the time of screening.

   * BMI = Weight(kg)/ Height(m)2
3. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
4. Those who are eligible for clinical trials based on laboratory(hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
5. Those who agree to contraception during the participation of clinical trial.
6. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those with clinically significant diseases or history in digestive systems, cardiovascular system, endocrine system, respiratory system, blood/tumor, infectious disease, kidney and urogenesis system, mental/nervous system, musculoskeletal system, immune system, otolaryngology, skin system, ophthalmology system, etc.
2. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
3. Those who have used drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, within 1 month before the first dosing date, or who have used drugs that may interfere with this study within 10 days before the first dosing day (However, clinical investigational drugs) Participation is possible in consideration of pharmacokinetic and pharmacodynamic characteristics such as interaction with concomitant drugs and half-life of concomitant drugs)
4. Those who have participated in other clinical trials or bioequivalence studies within 6 months of the first administration date and administered the investigational drug
5. Those who donated whole blood within 8 weeks of the first dose, or donated component blood within 2 weeks, or received blood transfusion within 4 weeks
6. Those who meet the following conditions within 1 month of the first administration date

   * In the case of men, alcohol consumption in excess of 21 drinks/week on average
   * For women, alcohol consumption in excess of 14 drinks/week on average

     (1 glass = 50 mL of soju or 30 mL of Western liquor or 250 mL of beer)
   * Smoking in excess of 20 cigarettes per day on average
7. A person who falls under any of the following

   * Patients with hypersensitivity to this drug or any of its components
   * Because this drug contains lactose, patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
8. Persons who are judged unsuitable for participation in this clinical trial by the principal investigator (or the authorized study doctor) for reasons other than the above selection/exclusion criteria
9. In the case of female volunteers, those who are pregnant or suspected of being pregnant or are lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-388, D418 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72 hours
  Area under the CKD-388/D418 concentration in blood-time curve from zero to final
Cmax of CKD-388, D418 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72 hours
  The maximum CKD-388/D418 concentration in blood sampling time

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, Principal Investigator — South Korea
Locations (1):
- H plus Yangji hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No